CLINICAL TRIAL: NCT03032926
Title: Enhancing Specificity and Predictability of CBT Outcome for Pediatric Anxiety Disorders: A Pilot Test of a Potential Biomarker for Treatment Response Across Development
Brief Title: A Pilot Study of Fear Extinction Learning in Anxious Youth
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1310014441
Record Dates: First submitted 2017-01-23; First posted 2017-01-26 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Anxiety Disorder of Childhood
Keywords: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open Trial: N/A - Open Trial
  Interventions: Behavioral: Open Trial

INTERVENTIONS:
Behavioral: Open Trial — Behavioral Intervention

SUMMARY:
The goal of this proposed study is to identify a potential biobehavioral marker of CBT outcome in the most common child and adolescent anxiety disorders, including separation anxiety disorder (SAD), social phobia (SoP), and generalized anxiety disorder (GAD), and to replicate in a clinical sample the previous finding from animal and non-clinical human samples that a difference exists in extinction learning across development.

DETAILED DESCRIPTION:
Study Sample and Design: The study will utilize an open treatment pilot trial design. Participants will include 10 individuals, ages 11-18, with a primary anxiety disorder diagnosis. Participants must not have failed prior trials of CBT. Participants on psychiatric medication must be on a stable dose for at least 2 months prior to study participation and remain symptomatic to the level identified for study inclusion (ADIS CSR ≥ 4).

Measures: Independent evaluators will administer a comprehensive assessment at baseline and post-treatment. The Anxiety Disorder Interview Schedule for Children for DSM-5 (ADIS-C-5)19 will measure the primary outcome of change in clinical severity of anxiety disorder symptoms across age groups. The Clinical Global Impression Scale (CGI) will assess overall symptom severity. The PARS and the MASC will provide secondary, dimensional measures of anxiety. In addition, we will measure treatment adherence and parent engagement as important secondary variables.

Fear Conditioning & Extinction Paradigm: Subjects will participate in a laboratory test of extinction training prior to CBT in order to establish extinction learning as a potential predictive marker of treatment outcome. Subjects will be exposed to two shapes on a computer screen, one shape (conditioned stimulus (CS+) will be paired with an aversive sound (unconditioned stimulus) on 38% of the trials, whereas the other shape will never be paired with aversive sound (CS-)20. A day later, individuals will undergo extinction training in which the two conditioned stimuli will be repeatedly presented without the unconditioned stimulus. Extinction will be measured as the difference score of skin conductance response to the CS+ and CS-.

Exposure Therapy Intervention: investigators will offer participants an 8 session exposure therapy intervention. Session one will consist of psychoeducation and completion of an exposure hierarchy. Sessions 2-7 will consist of weekly gradual exposure sessions. Session 8 will include review, relapse prevention and referral to additional treatment if needed. Assessment measures will be given at the completion of each exposure session to assess individual differences in symptom change related to exposure therapy. All treatment sessions will be videotaped to ensure fidelity to treatment manual and modules.

Data analysis plan: Investigators will track the monthly number of participants screened and enrolled to determine feasibility of a larger trial, as well as session attendance, study attrition, treatment adherence and patient safety to assess acceptability of the selected measures and interventions. Though this pilot will not be adequately powered to detect statistical significance, the investigators will execute a preliminary test of the association between performance on the extinction learning task and treatment outcome, and the investigators will assess age group differences in extinction learning and treatment outcome to determine early proof of concept.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7-25 years inclusively (i.e., must be at least 7 years) at the point of consent
* Primary DSM 5 diagnosis of SepAD, SocAD, OCD, specific phobia, or panic disorder on the ADIS-IV-C/P
* Anxiety severity of moderate or greater (CGI-S >3 and functional impairment (CGAS score 60)

Exclusion Criteria:

* Estimated child Full Scale IQ < 80, as measured by the vocabulary and block design subtests of the WISC-III) (Gate B). If a potential subject has a verified IQ score in the three years prior to enrollment as measured by the WISC-III, IIIR, K-ABC, or Stanford-Binet no IQ assessment is required.
* Child meets criteria for current primary or co-primary major depressive disorder, conduct disorder or substance abuse
* Child meets criteria for Major Depressive Disorder at greater severity than anxiety disorder (Gate B)
* Subjects with the following lifetime psychiatric disorders will be excluded: bipolar disorder, PDD (Asperger's, autism), MDD with psychosis, schizophrenia, and schizoaffective disorder
* Current use of psychotropic medication or clinical indication for use of psychotropic medication (except for youth entering on a stable psychostimulant regimen for ADHD)
* Recent treatment with psychotropic medication within 6 weeks of study entry for fluoxetine, within 2 weeks for other SSRIs, and within 4 weeks for neuroleptics (Gates A, B).
* Child has failed an adequate trial of CBT for anxiety within the previous 2 years (at least 10 treatment sessions over a period of less than 1 year conducted by a licensed provider of CBT)
* Child has a major neurological disorder, a major medical illness or hearing impairment that requires a prohibited episodic or chronic systemic medication or that would interfere
* Child is pregnant as indicated by history or a positive pregnancy test at Gate B. Sexually active girls must agree to use an effective form of birth control, either hormonal (BCP, Depo-Provera or Norplant), spermicide (foam or vaginal suppository) or a barrier method (condoms, diaphragm, cervical cap) or a combination of barrier/spermicide contraception in order to participate in the study.
* Child poses a significant risk for dangerousness to self or to others
* Child or parent is non-English speaking (unable to complete measures, IE ratings or treatment without the assistance of a translator) NYSPI and UCLA may recruit Spanish speaking subjects.
* Child is a victim of ongoing or previously undisclosed child abuse requiring new department of social service report or ongoing department of social service supervision
* Child, for any reason, has missed more than 50% of school days in the 2 months preceding randomization. Home schooling does not require exclusion from the study under this exclusion criterion. Ambiguous cases are referred to Caseness Panel to avoid truncating the severity range differently across sites
* Child has a history of seizures

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Youth with anxiety disorders ages 7-25
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
ADIS Evaluation | 1 year
  Anxiety Disorders Interview Schedule for DSM-5-Adult Version

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Bennett, PhD, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No